CLINICAL TRIAL: NCT06851520
Title: Retrospective Analysis of Different Quadratus Lumborum Block Techniques on Recovery Quality and Analgesic Consumption in Radical Cystectomy Patients
Acronym: QLB-CYS
Status: Completed | Type: Observational
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Onur Baran, Assistant Professor, Namik Kemal University
Other Study IDs: 2024.297.11.04
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Bladder Cancer; Postoperative Pain Management; Opioid Consumption; Recovery Quality
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Anterior QLB Group: Patients who underwent radical cystectomy under general anesthesia and received anterior quadratus lumborum block (QLB) for postoperative analgesia.
  Interventions: Procedure: Anterior Quadratus Lumborum Block (QLB)
- Posterior QLB Group: Patients who underwent radical cystectomy under general anesthesia and received posterior quadratus lumborum block (QLB) for postoperative analgesia.
  Interventions: Procedure: Posterior Quadratus Lumborum Block (QLB)

INTERVENTIONS:
Procedure: Anterior Quadratus Lumborum Block (QLB) — A regional anesthesia technique where local anesthetic is injected anterior to the quadratus lumborum muscle under ultrasound guidance for postoperative pain management.
  Groups: Anterior QLB Group
Procedure: Posterior Quadratus Lumborum Block (QLB) — A regional anesthesia technique where local anesthetic is injected posterior to the quadratus lumborum muscle under ultrasound guidance for postoperative pain management.
  Groups: Posterior QLB Group

SUMMARY:
This retrospective observational study evaluates the effects of different Quadratus Lumborum Block (QLB) techniques on postoperative recovery and total opioid consumption in patients undergoing radical cystectomy under general anesthesia. The study will analyze intraoperative and postoperative patient records from October 15, 2023, to October 15, 2024, at Tekirdağ Namık Kemal University Hospital.

Patients who received anterior or posterior QLB for postoperative analgesia will be included. Data collection will involve demographic information, total opioid consumption (morphine milligram equivalents), recovery quality scores (QoR-15), postoperative pain scores (Visual Analog Scale, VAS), time to first rescue analgesic administration, frequency of rescue analgesic use, and incidence of postoperative nausea and vomiting (PONV).

The retrospective analysis will compare the two QLB techniques to determine if there is a significant difference in postoperative opioid consumption and recovery quality. Statistical methods will be used to assess pain scores over time, opioid consumption, and overall recovery quality.

DETAILED DESCRIPTION:
Postoperative pain management plays a crucial role in optimizing recovery after radical cystectomy, as inadequate pain control can lead to increased opioid consumption and delayed rehabilitation. This retrospective observational study examines the effects of two different Quadratus Lumborum Block (QLB) techniques-anterior and posterior approaches-on postoperative pain and opioid consumption.

The study includes patients who underwent radical cystectomy under general anesthesia at Tekirdağ Namık Kemal University Hospital between October 15, 2023, and October 15, 2024. The primary focus is to compare total opioid consumption (morphine milligram equivalents) within the first 24 hours after surgery between the two groups.

Secondary outcomes include:

* Pain scores at multiple time points (0, 2, 6, 12, 24 hours), measured using the Visual Analog Scale (VAS)
* Postoperative recovery quality scores (QoR-15)
* Time to first rescue analgesic administration
* Frequency of rescue analgesic use
* Incidence of postoperative nausea and vomiting (PONV)

Data will be collected from intraoperative and postoperative patient records. Statistical analysis will compare anterior vs. posterior QLB techniques, evaluating differences in postoperative opioid consumption, pain relief efficacy, and recovery quality (QoR-15 scores).

This study aims to provide evidence-based insights into the use of regional anesthesia techniques for radical cystectomy patients, supporting the refinement of multimodal analgesia strategies to optimize pain management and minimize opioid exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent radical cystectomy under general anesthesia between October 15, 2023, and October 15, 2024.
2. Patients who received anterior or posterior quadratus lumborum block (QLB) for postoperative analgesia.
3. Age: 18-65 years.
4. ASA Physical Status Classification: I-III.
5. BMI < 35 kg/m².
6. Complete medical records available for retrospective review.

Exclusion Criteria:

1. Patients who received a different postoperative analgesia technique (e.g., epidural, TAP block).
2. Incomplete or missing medical records.
3. Psychiatric disorders that could affect pain perception and reporting.
4. Coagulopathy or bleeding disorders.
5. Hepatic or renal failure.
6. Chronic opioid use before surgery.
7. Patients who required unplanned conversion to open surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients (18-65 years old) who underwent radical cystectomy under general anesthesia at Tekirdağ Namık Kemal University Hospital between October 15, 2023, and October 15, 2024. Patients were retrospectively selected based on the administration of anterior or posterior Quadratus Lumborum Block (QLB) for postoperative analgesia. Patients with complete medical records were included, while those with missing data, coagulopathy, chronic opioid use, or unplanned open surgery conversion were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Total Opioid Consumption (Morphine Milligram Equivalents) in the First 24 Hours | 0-24 hours postoperatively
  The total amount of opioids (converted to morphine milligram equivalents) administered postoperatively within the first 24 hours following radical cystectomy.
  Continuous variable (mg of morphine equivalent)

SECONDARY OUTCOMES:
Pain Scores Using Visual Analog Scale (VAS) at Multiple Time Points | 0, 2, 6, 12, and 24 hours postoperatively
  Postoperative pain levels measured using the Visual Analog Scale (VAS) at predetermined time points: 0, 2, 6, 12, and 24 hours.
  Ordinal variable (0-10 VAS score, higher scores indicate more pain)
Postoperative Recovery Quality (QoR-15 Score) | 24 hours postoperatively
  Recovery quality assessed using the QoR-15 questionnaire, a validated patient-reported outcome measure.
  Continuous variable (QoR-15 total score, higher scores indicate better recovery quality)
Time to First Rescue Analgesic Administration | 0-24 hours postoperatively
  The duration (in minutes) from the end of surgery until the first administration of rescue analgesia.
  Continuous variable (minutes)
Frequency of Rescue Analgesic Use | 0-24 hours postoperatively
  The number of times rescue analgesics were administered during the first 24 hours postoperatively.
  Count variable (number of doses)
Incidence of Postoperative Nausea and Vomiting (PONV) | 0-24 hours postoperatively
  The proportion of patients who experience postoperative nausea and vomiting within the first 24 hours.
  Binary variable (Yes/No; presence of PONV)

CONTACTS AND LOCATIONS:
Locations (1):
- Tekirdağ Namık Kemal University Hospital, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korgvee A, Veskimae E, Huhtala H, Koskinen H, Tammela T, Junttila E, Kalliomaki ML. Posterior quadratus lumborum block versus epidural analgesia for postoperative pain management after open radical cystectomy: A randomized clinical trial. Acta Anaesthesiol Scand. 2023 Mar;67(3):347-355. doi: 10.1111/aas.14188. Epub 2023 Jan 3. PMID 36547262